CLINICAL TRIAL: NCT03782909
Title: Evaluation of a Behavioural Intervention Using App Technology in Cystic Fibrosis
Brief Title: Evaluation of a Behavioural Intervention Using App Technology in CF
Acronym: EAT-CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STH20240
Record Dates: First submitted 2018-12-17; First posted 2018-12-20 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Cystic Fibrosis
Keywords: Nutrition; Weight; BMI; Behaviour change
MeSH Terms: conditions — Cystic Fibrosis; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behaviour change intervention (Experimental): Intensive behaviour change for 6 weeks, followed by a maintenance phase for 6 weeks
  Interventions: Behavioral: Behaviour change intervention

INTERVENTIONS:
Behavioral: Behaviour change intervention — The behaviour change intervention consists of;
  1. Feedback via an app based food diary
  2. Coaching with problem solving and implementation plans
  The intensive phase consists of 2 home visits and 4 phone calls and the use of the app The maintenance phase consists of use of the app if the PWCF wishes to continue using it

SUMMARY:
Cystic Fibrosis (CF) is a lifelong condition which causes the lungs and digestive system to become clogged with thick, sticky mucus. This leads to recurrent chest infections and reduced nutrient absorption from food. The average age at death is 31 years, usually from respiratory failure. The nutritional status of people with CF (PWCF) is important to help them live healthier and longer.

It is recommended that adults with CF achieve a BMI of 23 for males and 22 for females. However, fewer than 50% of adults with CF achieved that target BMI despite effective nutritional support to help weight gain. There is a clear need for a behavioural intervention that can help PWCF use the available nutritional support.

This is a feasibility study to try out a multi-component behavioural intervention supported by a nutrition app. The intervention is designed to help PWCF use their nutritional support to gain weight. It will focus on testing the methods and procedures to be used on a larger scale, improving the behavioural intervention and estimating how many people are needed for the larger trial.

Eligible patients will be invited to participate, and the investigators anticipate recruiting 6 participants. The participants will have 6 weeks of intensive intervention, which will include a mix of clinic visits, home visits and telephone calls followed by 6 weeks of maintenance phase. Data will be collected during clinic visits at baseline, week 6 and week 12 along with weight monitoring at home.

The investigators will interview each participant at the end of the study period to improve the intervention and study processes based on participant feedback.

The investigators hypothesised that using a nutrition app, along with regular input from a dietitian, will help PWCF to use the available nutritional support.

ELIGIBILITY:
Inclusion Criteria:

* adult people with CF looked after at the Sheffield Adult CF Centre
* best BMI of <23 for males and <22 for females between June 2018 and November 2018

Exclusion Criteria:

* patients in palliative phase of disease
* patients who are pregnant
* patients who have no capacity to consent to participate in the study
* patients who are unable to communicate by telephone for coaching

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who accepted invitation to participate as a marker of feasibility | 4 weeks

SECONDARY OUTCOMES:
Participants' opinion about the behavioural intervention | 3 months
  A semi-structured interview will be used for thematic analysis
Participant attrition rate and phases of the study whereby the attrition occurs | 3 months
Participants' opinion about the study processes | 3 months
  A semi-structured interview will be used for thematic analysis
Participants' suggestions for further improvement of the intervention and study processes | 3 months
  A semi-structured interview will be used for thematic analysis
Proportion of adults who fulfils the BMI criteria for recruitment with IT facilities | 4 weeks
Resources (time) needed by the investigators to deliver the intervention | 3 months
  Time will be used as a measurement tool to quantify total time required to deliver the intervention
Proportion of days with missing nutritional data, as a marker of feasibility | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Hallamshire Hospital, Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom